**Title:** The Andrews Return to Sport ACL Score: A Developmental Study

**Principal Investigator:** Adam Anz, M.D.

**Co-Investigators:** James Andrews, M.D.

Steve Jordan, M.D.

Roger Ostrander, M.D.

Tyler Opitz, DPT, SCS, CSCS

Albi Gilmer, MSPT, OCS

Ron Courson, ATC, PT, NRAEMT, CSCS

Jessi Truett, MA, BCBA

Joshua Cook, B.S.

Chandler Bridges, M.S.

Thomas Denney Jr., Ph.D.

Funding Mechanism: Florida State Grant

**Institution:** Andrews Institute

1020 Gulf Breeze Pkwy.

Gulf Breeze, FL 32561

(850) 916- 8590

Version: 1.0

## **Table of Contents**

| Abbreviations and Definitions | 4 |
|-----------------------------------|----|
| Background / Scientific Rationale | 5 |
| Objective: | 7 |
| Protocol Design | 7 |
| Hypotheses | 7 |
| Alternative Hypothesis: | 8 |
| Null Hypothesis: | 8 |
| Treatment Plan | 8 |
| Return To Sport Assessments: | 11 |
| Isokinetic Strength Testing: | 11 |
| Magnetic Resonance Imaging | 11 |
| Functional Movement Assessments: | 12 |
| Single Leg Squats: | 12 |
| Jump Analysis: | 13 |
| Single Leg Press: | 14 |
| Back Squat | 14 |
| Y Balance Test (YBT) | 14 |
| Patient Reported Outcomes | 15 |
| Tampa Kinesiophobia Scale: | 16 |
| Sports Participation Assessment: | 16 |

| Reinjury Assessment: | 16 |
|---|---|
| International Knee Documentation Committee Subjective Knee Evaluation Form (IKDC): | 17 |
| Patient Reported Outcomes Measurements Information Systems (PROMIS) | 17 |
| Single Assessment Numeric Evaluation (SANE) | 17 |
| Review of Safety | 18 |
| Adverse Event (AE) | 18 |
| Serious Adverse Event (SAE) | 18 |
| Unanticipated Problem (UP): | 18 |
| AE & SAE Collection and Reporting | 19 |
| Risks and Discomforts | 20 |
| Safety Monitoring Plan | 20 |
| Quality Control and Assurance | 20 |
| Regulatory Requirements | 20 |
| 21 CFR 50- informed consent: | 20 |
| Consent Withdrawal: | 21 |
| Participant Confidentiality | 21 |
| Data Analysis & Management Procedures | 22 |
| Data Collection | 22 |
| Statistical Analysis | 22 |
| References | 23 |
| Appendix | 25 |

# **Abbreviations and Definitions**

| ACL | Anterior cruciate ligament | JHFT | Jump Height by Flight Time |
|---|---|---|---|
| AE | Adverse Event | MRI | Magnetic resonance imaging |
| AREF | Andrews Research and Education | OKC | Open Kinetic Chain |
| Found | ation | PI | Principal Investigator |
| CRF | Case Report Form | PRO | Patient Reported Outcomes |
| DHHS<br>Service | S Department of Health and Human | RTP | Return to Play |
| EDC | Electronic Data Capture | RTS | Return to Sport |
| FMS | Functional Movement Screening | QA | Quality Assurance |
| GCP | Good Clinical Practice | SAE | Severe Adverse Event |
| HIPA | A Health Insurance Portability and | SOC | Standard of Care |
| | entability Act | SOP | Standard Operating Procedure |
| $H_0$ | Null Hypothesis | TSK | Tampa Scale for Kinesiophobia |
| $H_1$ | Alternative Hypothesis | YBT | Y Balance Test |
| IRB | Institutional Review Board | | |


**Background / Scientific Rationale** 

It is estimated that 250,000 anterior cruciate ligament (ACL) injuries occur in the United States

per year (Griffin et al., 2000, Gianotti et al., 2009). With ACL injuries being one of the most

frequent injuries in both contact and noncontact sports, medical professionals need reliable tools

to treat injured athletes and return them to sport in a safe/timely fashion (Harris et al., 2013).

Along with the prevalence of initial injury, reinjury rates may be up to 30% in young active

patients who undergo ACL surgical interventions. With the rate of return to competitive play

post-ACL injury being 55%, it is imperative to create a systematic quantitative algorithm to

safely return athletes to competitive play after ACL injury (Ardner et al., 2014). In addition to the

primary injury often there is additional concern for instability of the knee, increased joint laxity,

reduced activity and participation, as well as an increased risk of knee osteoarthritis in the future

for the athlete (Lohmandeder et al., 2004). Along with the play time missed for the athletes, ACL

injuries are associated with significant physical and mental harm as well as a lower health-related

quality of life which supports the need for effective Return to Sport assessments. However, the

current literature is limited regarding the standardization and data-driven decision in regards to

return-to-sport algorithms (Creighton et al., 2010). Return-to-sport algorithms require further

development.

Regenerative medicine technologies have the potential to expedite return to sport times after

injury and surgery. However, to objectively study the application of regenerative medicine

technologies to ACL injury and surgery, the development of an objective measurement system

for the safe and appropriate return of patients to sport is required. Ensuring patients are being

safely returned to their sports after treatments for ACL injuries is important to decrease the risk

of reinjury. As noted in Grindem et al. (2016), athletes returning to sport with asymmetrical


Version Date: 10NOV2021

quadricep strength have a significant risk increase for reinjury. After sustaining injury and operative intervention, a systematic evaluation process is needed to evaluate athletes' progress towards returning to sport. To safely return to sport, an athlete must restore range of motion, strength, and stability and control across the affected and unaffected knee (Wilk et al., 2012; Bodor, 2001). With current advancements in technology, an up-to-date quantitative return to sport algorithm is presented. Multiple measures are required to capture the risk factors for reinjury such as imbalances and weaknesses that are not always evident in observation. The purpose of this study is to develop the Andrews ACL S.C.O.R.E (Subjective Clinical Outcome Return to Play Evaluation.) Development will begin with baseline measures and re-evaluation during the rehabilitation progression to address asymmetries and movement inefficiencies in a data driven manner with the ultimate goal of returning to play safely, without reinjury. A modern return to sport algorithm will include patient reported outcome measures, objective/modern strength and ability testing, and MRI evaluation of the reconstructed ACL tissue. Ardern et al. (2014) report the importance of assessing the psychological factors that impede athletes from returning to sport after ACL reconstruction. To address these individualized factors, patient reported outcomes are used to quantify these measures.

A comprehensive assessment is required to ensure an athlete's ability to safely return to sport is identified. This Return to Sport assessment must incorporate the overall health of the individual and assess specific measures of the affected ACL area. These qualities of assessment include the need for their strength to be at or near their preinjury level with symmetry to the non-injured leg, range of motion at or near their preinjury level with symmetry to the non-injured leg, joint stability at or near their preinjury level with symmetry to the non-injured level and confidence in movement comparable to the confidence in movement to the non-injured leg. As found by


Ardern et al. (2014) symmetry hopping in movement has positive predictive factors for returning

to competitive sport levels after ACL reconstruction. The functional movement screening

assessment, a low-cost assessment, is also widely used to assess current functioning level. This

assessment includes seven movement patterns to ensure the whole-body biomechanics can be

assessed. The FMS assessment will provide a quantitative assessment of functional movement

**Objective:** 

This project will develop a data driven decision making model to assess a competitive athlete's

readiness to return to sport after ACL injury and surgery safely. A specific audience and return to

activity level specification is required for complete return to sport studies (Gokeler et al., 2017).

This Return to Sport algorithm is targeting competitive pre-collegiate and collegiate athletes with

a return to sport that is congruent with their pre-injury level of play.

Return to Sport-Obtaining medical clearance to participate in competitive sports at the athlete's

pre-injury level

Safely- Returning to pre-injury competitive level without instances of reinjury of the same ACL

**Protocol Design** 

This will be a prospective cohort study of 100 competitive level pre-collegiate and collegiate

level athletes who have sustained an ACL injury requiring reconstruction with a length of

enrollment of 36 months.

**Hypotheses** 


**Alternative Hypothesis:** 

The prospective capture of multimodal data will improve the safe return of athletes to sport after

ACL surgery and allow for the evaluation of regenerative medicine technologies to improve this

process.

Patient reported outcomes and return to sport times will correlate directly with MRI objective

scores and biometric strength/movement scores.

**Null Hypothesis:** 

The prospective capture of multimodal data will not show improvement in the rate of safe return

of athletes to sport after ACL surgery.

Patient reported outcomes and return to sport times will not directly correlate with MRI

objective scores and biometric strength/movement scores.

**Treatment Plan** 

For the one hundred participants recruited for this study, the duration of the treatment plan will

be 24 months. Each of the participants will be qualified for the study due to falling within all

inclusion criterion and no exclusion criterion. The screening of the inclusion criterion will occur

at visit one of the study. At this time, the AREF Research Team will review and collect informed

consent from each participant. Visit two will occur three (3) months after each participant's ACL

reconstruction surgery. At this time, an evaluation by the treating physician will occur along

with functional movement assessment and MRI. Visit three will occur six (6) months after each

participant's ACL reconstruction surgery. At this time, an evaluation by the treating physician


will occur along with functional movement assessment and MRI. Visit four will occur nine (9)

months after each participant's ACL reconstruction surgery. At this time, an evaluation by the

treating physician will occur along with functional movement assessment and MRI. Visit five

will occur twelve (12) months after each participant's ACL reconstruction surgery. At this time,

an evaluation by the treating physician will occur along with functional movement assessment

and MRI. Visit six will occur eighteen (18) months after each participant's ACL reconstruction

surgery. At this time, an evaluation by the treating physician will occur along with functional

movement assessment and MRI. Visit seven will occur twenty-four (24) months after each

participant's ACL reconstruction surgery. At this time, an evaluation by the treating physician

will occur along with functional movement assessment and MRI. At each time point, the treating

physician or the therapist performing the functional movement assessment can choose to limit

the functional movement assessment if there are concerns that the patient may not be ready for

the expected load of one or more elements of the functional movement assessment.

At each monthly time point after ACL reconstruction patient reported outcomes will be collected

by the research team to assist in assessing the overall health and confidence in Return to Sport

for each athlete. The following patient reported outcomes will be collected in written or

electronic format after informed consent has been obtained from each participant: Sports

Participation, Reinjury, Tampa Kinesiophobia Scale, IKDC, PROMIS, SANE.

**Participation:** 

A total of 100 competitive pre-collegiate or collegiate athletes will be recruited for participation

in the Andrews Return to Sport algorithm study. Participants in the study will be individuals who

have provided informed consent to the research team to adhere to the provided research protocol.


**Inclusion Criterion:** 

One hundred (100) pre-collegiate or collegiate level athletes will be included in this study. They

will fall within the following inclusion criterion:

1. Age 14-24 years

2. Require ACL reconstruction surgery

3. No other ligament injury which would require repair or reconstruction to lower extremity

is present as assessed by treating physician

4. Exhibits desire to return to pre-injury competitive level

5. Assessed to be in good physical health condition by the treating physician

**Exclusion Criterion:** 

1. Requires more than one ACL reconstruction surgery at time of screening

2. Has comorbid lower extremity diagnoses which would impede return to sport as assessed

by the treating physician

3. Does not desire to return to pre-injury competitive sport level

**Benefits:** 

Each study participant will be provided with a total five hundred dollars (\$500.00) for their

participation in the study through the 24-month period. The \$500.00 will be dispersed on the

following predetermined schedule. \$100.00 at Visit 2, \$100.00 at Visit 3, \$100.00 at Visit 5,

\$100.00 at Visit 6, and \$100.00 at Visit 7. If a participant withdraws from the study the


monetary benefits will not be dispersed after the withdrawal date. However, there will be no

effect on the medical care provided if a participant withdraws from the study.

**Return To Sport Assessments:** 

**Isokinetic Strength Testing:** 

Isokinetic strength testing is crucial to assess the muscular strength of the quadricep and

hamstring after ACL reconstruction. Due to the high rate of reinjury with known predictive

factors due to imbalance in strength, a quantitative measure of balance of strength is required to

guide return to sport decision making. An isokinetic dynamometer will be used to assess knee

extensor and flexor strength (Riesterer et al., 2020). Isokinetic strength testing will support the

Andrews Return to Sport algorithm through multimodal functional assessments.

**Magnetic Resonance Imaging** 

Magnetic Resonance Imaging (MRI) will be used as a noninvasive assessment tool to obtain

quantitative measures to assess progress in graft maturity and rehabilitation towards safe return

to sport. As the injured ACL undergoes ligamentization, MRI will be used to monitor the

progress of each participant through T2\* analysis and volume at the following time intervals:

3months, 6months, 9months, 12months, 18months, and 24months. MRIs will review the

integrity of each graft, placement within the tunnel, and tunnel healing, and healing of the donor

site (Grassi et al., 2016).


**Functional Movement Assessments:** 

The functional movement screening assessment (FMS) is widely used to assess current

functioning level and does not require significant monetary resources to provide this assessment.

This assessment includes seven movement patterns to ensure the whole-body biomechanics can

be assessed. The movements required are deep squat, hurdle step, inline lunge, shoulder

mobility, active straight leg raise, trunk stability push up, and rotary stability assessment. FMS

screening will be used to identify the precursor deficits which could lead to reinjury. These

deficits include increased anterior tibial shear force, decrease knee flexion, decreased hip flexion,

increased knee internal rotation, increased trunk flexion, and increased lumbar hyperextension.

The FMS assessment will provide a quantitative assessment of functional movement on a 0-3

scale as follows (Hoogenboom, Voight, Cook, & Rose, 2013).

3- Individual can perform the movement without any compensation.

2- Individual can perform the movement but must utilize poor mechanics and compensatory

patterns to accomplish the movement.

1- One is given if the individual cannot perform the movement pattern even with compensation.

0- Individual reports pain during activity.

**Single Leg Squats:** 

The single leg squat assessment is commonly used to evaluate the eccentric and concentric

contractions of the muscles in the upper leg, lower leg, and hip (Bailey et al., 2010). This test

was first executed and defined the method for performing by Livengood (2004) to assess

balance, strength, and the kinetic chain. To rate the single leg squat test, Livengood also assigned


a scale to the test (Figure 1). Each participant will be instructed to squat down to approximately

60 degrees with a time constraint of six seconds while holding one leg suspended in the air.

When analyzing the movements within the single leg squat, researchers assess the functioning

and symmetry of following muscles and the activity associated: vastus medialis obliquus, gluteus

medius, hip flexion, hip abduction, and knee flexion (Table 1).

Jump Analysis:

The jump analysis highlights the importance of the monthly psychological data review

completed by the Kinesiophobia Scale. In review of this data, the psychological apprehension

will guide the functional jump analysis. The jump analysis will occur initially from both legs to

address psychological apprehension (Davies et al., 2017). From this assessment, calculation is

made based on the allometric scaling to each participant's height (Davies et al., 2017).

Additionally, flight time will be measured as defined by the time (s) when the participant's feet

leave the platform and subsequently contact the platform again (Jordan et al., 2020).

Additionally, the jump height by flight time (JHFT) will be measured. JHFT is defined as the

distance the marker on the malleolus moved from lowest point when in contact with the platform

to the highest point during the jump.

A single leg hop assessment will also be performed across both the injured and non-injured legs.

The score for this assessment is the distance travelled from the start to the location of the

posterior heel of the landing leg (Manske & Reiman, 2013). The variability of scores across the

injured and non-injured leg will be used as a measure of symmetry in function movement for

each athlete.


Additionally, a double leg hop will be scored during the jump analysis. The score for this

assessment is the distance travelled from the start to the location of the posterior heel of the

landing leg (Manske & Reiman, 2013). Additionally the participant's jump will be assessment

for symmetry in takeoff and landing across both the injured and uninjured leg.

**Single Leg Press:** 

Additional readiness measures will be assessed through the single leg press motion. As the

participants progress in rehabilitation a body weight single leg press will be completed across

both the injured and non-injured leg until failure. Then a single leg press with 25% body weight

will be completed until failure. This measure of repetitions until failure will be used to assess the

current fatigue level of the injured leg regarding readiness to Return to Sport. This measure will

also occur quantitative data as a measure of deficit which will align with future reinjury rates.

**Back Squat** 

Each participant will undergo a back squat assessment as they progress in rehabilitation. Once

the investigator deems the participant stable in the descending, stable hold position, and

ascending motion. Each participant's movement pattern while completing a back squat will be

assessed for stability and strength in maintaining position.

Y Balance Test (YBT)

The Y Balance Test is a reliable, yet simple assessment to measure the participant's strength,

stability, balance, and confidence while moving in three different directions. The YBT requires

the participant to balance on one leg at a time and to reach as far as possible with the suspended

leg in three separate directions, anterior, posterolateral, and posteromedial. This assessment will


measure the level of rehabilitation by measuring the knee flexor and hip adductor strength after

ACL injury (Walker, 2016).

The test will follow the procedural order of:

1. Right Anterior

2. Left Anterior

3. Right Posteromedial

4. Left Posteromedial

5. Right Posterolateral

6. Left Posterolateral

At the completion of the above sequence the following calculations will occur:

Absolute Reach Distance (cm)= (Reach 1 + Reach 2 + Reach 3)/3

Relative Reach Distance (%) = Absolute Reach Distance/Limb Length X 100

Composite Reach Distance (%) = Sum of the 3 Reach Directions/3 Times the Limb Length X

100

**Patient Reported Outcomes** 

Monthly assessments of each participant's patient reported outcomes will be used to quantify

physical and psychological aspects of rehabilitation after ACL reconstruction monthly after

informed consent has been obtained and surgery has occurred.


Tampa Kinesiophobia Scale:

The fear of reinjury can be a barrier to the rehabilitation of competitive athletes after

ACL reconstruction. To operationalize the fear associated with reinjury the Tampa

Kinesiophobia (TSK) will be provided monthly to participants in the study to complete

(Lundberg et al., 2009). Kinesiophobia is defined as the fear of movement (Lundberg et

al., 2009). This measure will be collected to evaluate progression in rehabilitation to take

into account not only the physical health of the injured athlete but also the psychological

effects and rehabilitation.

**Sports Participation Assessment:** 

A sports participation assessment will be completed monthly by the participants of the

research project to quantify the participant's participation in sports activity during the

rehabilitation period.

**Reinjury Assessment:** 

A monthly injury questionnaire will be provided to each participant of the study to assess

the rate of reinjury during the rehabilitation process. If reinjury is noted in the monthly

questionnaire, the AREF research team will alert the principal investigator to ensure

continuity of care is provided.


**International Knee Documentation Committee Subjective Knee Evaluation Form** 

(IKDC):

The International Knee Documentation Committee Subjective Knee Evaluation (IKDC)

form will contribute to the comprehensive data set to evaluate each participant's

confidence in performance on a monthly schedule. IKDC has 19 questions that will take

approximately 3-5 minutes for each participant to complete monthly. IKDC data will be

collected by the AREF research team and reviewed with the primary investigator.

**Patient Reported Outcomes Measurements Information Systems (PROMIS)** 

The patient reported outcomes measurement information system (PROMIS) is a

measurement system used monthly in this project to assess monthly the overall health

functioning and rehabilitation levels of each participant (Brodke, Saltzman, & Brodke,

2016). AREF will collect this data and alert the primary investigator if any adverse

outcomes are found. The addition of the PROMIS data is required to ensure that a

comprehensive assessment of overall functioning is reviewed in the determination of

athlete readiness to return to sport.

**Single Assessment Numeric Evaluation (SANE)** 

The SANE assessment is a single question patient reported outcome from a rating of 0-

100 for each participant to score their current functioning in comparison to their pre-

injury functioning level (O'Connor & Ring, 2019). This assessment will be collected

monthly after ACL reconstruction by the AREF research team for each participant.


**Review of Safety** 

Adverse Event (AE)

An adverse event is any untoward or unfavorable medical occurrence in the human subject,

including any abnormal sign, symptom, or disease, temporally associated with the subject's

participation in the research, whether considered related to the subject's participation in the

research or not considered related to the subject's participation in the research.

Serious Adverse Event (SAE)

Serious adheres events are any events that:

• Result in death

• Is life threatening, or places the participant at immediate risk of death from the event as it

occurred

• Requires or prolongs hospitalization

• Causes persistent or significant disability or incapacity

• Results in congenital anomalies or birth defects

• Is another condition which investigators just to represent significant hazards

Unanticipated Problem (UP):

Defined by DHHS 45 CFR part 46 as any incident, experience, or outcome that meets the

following criteria.


unexpected, in terms of nature, severity, or frequency, given (a) the research procedures

that are described in the protocol-related documents, such as the IRB-approved research

protocol and informed consent document; and (b) the characteristics of the study

population.

• related or possibly related to participation in the research (in this guidance document,

possibly related means there is a reasonable possibility that the incident, experience, or

outcome may have been caused by the procedures involved in the research);

• suggests that the research places participants or others at a greater risk of harm (including

physical, psychological, economic, or social harm) than was previously known or

recognized.

AE & SAE Collection and Reporting

Throughout the study the research team will monitor the occurrence of AE and SAE. Data will

be collected if an instance occurs, and the PI will be notified. All AE data, such as onset date,

resolution date, outcome and treatments given will be documented in the source documents and

will be recorded in the EDC and analyzed for severity to follow reporting protocol if severity

level.

Follow-up will occur using the provided safety monitoring form if AE occurs. The follow up will

end either when the symptoms resolve or up to 30 days past the end of the study participation.


**Risks and Discomforts** 

As with any research involving participants, there is the inherent risk of a breach in patient

confidentiality though this will be minimized using participant code numbers and adherence to

all HIPAA guidelines.

**Safety Monitoring Plan** 

The safety of each participant will be monitored through multiple channels as the primary focus

on this project is to ensure the safe return to sport for each participant. Along with the medical

evaluation performed at each of the seven study visits. Monthly patient reported outcomes will

be collected and reviewed to ensure no additional injury or premature return to sport has

occurred. Any deviation from protocol recommendations will be reported by the AREF research

team to the principal investigator to assess and rectify participant actions if needed.

**Quality Control and Assurance** 

All protocols will be monitored and analyzed data will be checked for accuracy by the principal

investigator and /or a designated AREF research team member. All medical data will be kept in

compliance with HIPAA guidelines.

**Regulatory Requirements** 

21 CFR 50- informed consent:

In adherence to the 21 CFR 50, Protection of Human Subjects Guidelines, the informed consent

process will be performed by one of the study investigators or staff, in the research office on


paper or electronically via REDCap. REDCap is a secure web application for building and

managing online surveys and databases. While REDCap can be used to collect virtually any type

of data in any environment (including compliance with 21 CFR Part 11, FISMA, HIPAA, and

GDPR), it is specifically geared to support online and offline data capture for research studies

and operations. The REDCap Consortium, a vast support network of collaborators, is composed

of thousands of active institutional partners in over one hundred countries who utilize and

support their own individual REDCap systems. All participants will have the study described to

them and will be given as much time as they require to read an approved, IRB stamped version

of the informed consent document. The designee will review with each participant that they are

free to refuse to participate in the study or to withdraw from it at any time.

After physical or electronic signing of the informed consent document, participants will be given

a copy for their records. No aspects of the study will be conducted prior to obtaining informed

consent from each participant.

**Consent Withdrawal:** 

During the informed consent process, participants will be informed that if at any point during the

study, consent may be withdrawn. To withdraw consent, participants can request in writing to

withdraw HIPAA authorization and the research site will not use or provide any health

information to researchers. At this time, the link between the participant's health information

will be severed with the research team. This process for consent withdrawal will be reviewed

with each participant and identified barriers will be addressed at the time of informed consent.

**Participant Confidentiality** 


Signed consent forms for each subject will be de-identified by a coding system with the subject's

unique study identification system. Authorization to use each subject's personal health

information will be obtained during the informed consent procedure to adhere to the federal

Health Insurance Portability and Accountability Act (HIPAA). The consent will specifically

grant permission to use health information obtained as part of the presented study.

**Data Analysis & Management Procedures** 

This study is anticipated to take 2 years to complete after informed consent is obtained for each

participant. All data will be entered into REDCap. The investigators will meet at appropriate

intervals to evaluate and analyze the data.

**Data Collection** 

Data will be collected using the Electronic Data Capture (EDC) system. Reports of data will be

used by internal site monitors to ensure accuracy of data elements. Data will be kept secure to

reduce chances of breach of confidentiality. Data will also be de-identified as another

confidentiality best practice measure.

**Statistical Analysis** 

All patient data will be entered into EDC. The investigators will meet at appropriate intervals to

evaluate and analyze the data. All compiled data will be de-identified.


#### References

Ardern, C. L., Taylor, N. F., Feller, J. A., and Webster, K. E. (2014). Fifty-five per cent return to competitive sport following anterior cruciate ligament reconstruction surgery: an updated systematic review and meta-analysis including aspects of physical functioning and contextual factors. Br. J. Sports Med. 48, 1543–1552. doi: 10.1136/bjsports-2013-093398

Bodor M.: Quadriceps protects the anterior cruciate ligament. J of Ortho Research 2001; 19: 629-633.

Boyle, M. & Galway, B.(n.d.). Evidence-based Clinical Protocols: Anterior Cruciate Ligament Injury & Reconstruction. Biodex Medical Systems, Inc.

Brodke, D, Saltzman, C., Brodke, D.;(2016). PROMIS for Orthopaedic Outcomes Measurement. Journal of American Academy Orthopedic Surgery. 2016;24: 744-749

Creighton DW, Shrier I, Shultz R, Meeuwisse WH, Matheson GO. Return-to-play in sport: a decision-based model. Clin J Sport Med. 2010 Sep;20(5):379-85. doi: 10.1097/JSM.0b013e3181f3c0fe. PMID: 20818198.

Davies, G., McCarty, E., Provencher, M., & Manske, R., (2017). ACL return to Sport Guidelines and Criteria. Current Rev Muscholosklet Med. 2017 10:307-314. (doi:10.1007/s12178-017-9420-9)

Fitzgerald, G.K, Axe, M.J., & Snyder-Mackler, L. (2000). The efficacy of perturbation training in nonoperative anterior cruciate ligament rehabilitation programs for physically active individuals. Physical Therapy, 80 (2), 128–40.

Gianotti S.M., Marshall S.W., Hume P.A., et al: Incidence of anterior cruciate ligament injury and other knee ligament injuries: a national population-based study. J Sci Med Sport 2009; 12: 622-627.

Griffin L, Agel K, Albohm M, et al. Noncontact anterior cruciate ligament injuries: risk factors and prevention strategies. J Am Acad Orthop Surg. 2000;8:1410159

Grindem, H., Syner-Mackler, L., Mokesnes, H., Engebretsen, L., & Risbeg, M. (2016). Simple Decision Rules Can Reduce Reinjury Risk by 84% After ACEL Reconstruction: the Deleware-Oslo ACL Cohort Study. Br J Sports Med 2016;50:804–808. . doi:10.1136/bjsports-2016-096031

Gokeler, Al., Welling, W., Zaffagnini, S., Seil, R., & Padu, D. (2017). Development of a test battery to enhance safe return to sports after anterior cruciate ligament reconstruction. Ken Surg Sports Traumatol Arthoscop. 25: 192-199. DOI 10.1007/s00167-016-4246-3

Hoogenboom, B., Voight, M., Cook, G., & Rose, G. (2013). Functional Movement Assessment. P. 463-495.


Jordan, M., Morris, N., Lane, M., Barnert, J., MacGregor, K., Heard, M., Robinson, S., & Herzog, W. (2020). Monitoring the Return to Sport Transition After ACL Injury: An Alpine Ski Racing Case Study. Front. Sports Act. Living. 2. Doi: 10.3389/fspor.2020.00012

Lohmander L.S., Englund P.M., Dahl L.L., et al: The long-term consequence of anterior cruciate ligament and meniscus injuries: osteoarthritis. Am J Sports Med 2007; 35: 1756-1769.

Lundberg, Mari, et al. "On what patients does the Tampa Scale for Kinesiophobia fit?" Physiotherapy Theory and Practice, vol. 25, no. 7, 2009, pp. 495–506. <a href="https://www.researchgate.net/publication/38112716\_On\_what\_patients\_does\_the\_Tampa\_Scale\_for\_Kinesiophobia\_fit.">https://www.researchgate.net/publication/38112716\_On\_what\_patients\_does\_the\_Tampa\_Scale\_for\_Kinesiophobia\_fit.</a>

Manske, R. & Reiman, M. (2013). Functional Performance Testing for Power and Return to Sport. Athletic Training. Functional Testing in Human Performance. DOI: 10.1177/1941738113479925

Miller RP, Kori S, Todd D. The Tampa Scale: a measure of kinesiophobia. Clin J Pain. 1991;7(1):51–52.

O'Connor & Ring. (2019). Correlation of Single Assessment Numeric Evaluation (SANE) with other Patient Reported Outcome Measures (PROMs). Archives of Bone and Joint Surgery. 7(4): 303-306.

Oxefit.(2021). Introducing Oxefit's XP1: An Unparalleled Strength Training Product with Real-Time Performance Assessment. Press Release. Dallas (Apr. 7, 2021).

Riesterer, Mauch, Gehring, Ritzman, and Wenning (2020). Relationship between pre-and post-operative isokinetic strength after ACL reconstruction using hamstring autograft. BMC Sports Science, Medicine and Rehabilitation. 12:63.doi: https://doi.org/10.1186/s13102-020-00215-7

Walker, O.(2016). The Y Balance Test. Science for Sport. Retrieved: https://www.scienceforsport.com/y-balance-test/

Wilk K.E., Macrina L.C., Cain E.L., et al: Recent advances in the rehabilitation of anterior cruciate ligament injuries. J Ortho & Sports Phys Ther 2012; 42: 153-171.


### Appendix

#### **Treatment Schedule:**

- 1. Visit 1- Screening Visit (Informed Consent/Review Inclusion and Exclusion)
- 2. Visit 2- (3 mo after ACL Reconstruction)- \$100.00 to participant
  - a. Strength/Functional Testing with a Therapist, MRI
- 3. Visit 3- (6 mo after ACL Reconstruction)- \$100.00 to participant
  - a. Strength/Functional Testing with a Therapist, MRI
- 4. Visit 4- (9 mo after ACL Reconstruction)
  - a. Strength/Functional Testing with a Therapist, MRI
- 5. Visit 5- (12 mo after ACL Reconstruction)- \$100.00 to participant
  - a. Strength/Functional Testing with a Therapist, MRI
- 6. Visit 6- (18 mo after ACL Reconstruction)- \$100.00 to participant
  - a. Strength/Functional Testing with a Therapist, MRI
- 7. Visit 7- (24 mo after ACL Reconstruction)- \$100.00 to participant
  - a. Strength/Functional Testing with a Therapist, MRI

PRO: Monthly

1. Sports Participation (Monthly)


| 2. | Reinjury (Monthly) |
|---|---|
| 3. | Tampa Kinesiophobia Scale (Monthly) |
| 4. | IKDC (Monthly) |
| 5. | PROMIS (Monthly) |
| 6. | SANE (Monthly) |
| MRI: | 3mo, 6mo, 9mo, 12mo, 18mo, 24mo |
| 1. | Volume |
| 2. | Mean T2* Values |
| Streng | th/Functional Testing with a Therapist: 3mo, 6mo, 9mo, 12mo, 18mo, 24mo |
| 1. | Isokinetic Strength Testing |
| 2. | FMS- Functional Movement Screening |
| 3. | Y-Balance |
| 4. | Single Leg Hop |
| 5. | Single Leg Press with Body weight (number of reps), 25% body weight (number of reps) |

Version: 1.0 Version Date: 10NOV2021

## Tampa Scale for Kinesiophobia

(Miller, Kori and Todd 1991)

| 1 – Subligly disagle | strongly disagre | ee |
|----------------------|------------------|----|
|----------------------|------------------|----|

2 = disagree

3 = agree

4 = strongly agree

| 1. I'm afraid that I might injury myself if I exercise | 1 | 2 | 3 | 4 |
|---|---|---|---|---|
| 2. If I were to try to overcome it, my pain would increase | 1 | 2 | 3 | 4 |
| 3. My body is telling me I have something dangerously wrong | 1 | 2 | 3 | 4 |
| 4. My pain would probably be relieved if I were to exercise | 1 | 2 | 3 | 4 |
| 5. People aren't taking my medical condition seriously enough | 1 | 2 | 3 | 4 |
| 6. My accident has put my body at risk for the rest of my life | 1 | 2 | 3 | 4 |
| 7. Pain always means I have injured my body | 1 | 2 | 3 | 4 |
| 8. Just because something aggravates my pain does not mean it is dangerous | 1 | 2 | 3 | 4 |


| 9. I am afraid that I might injure myself accidentally | 1 | 2 | 3 | 4 |
|---|---|---|---|---|
| 10. Simply being careful that I do not make any unnecessary movements is the safest thing I can do to prevent my pain from worsening | 1 | 2 | 3 | 4 |
| 11. I wouldn't have this much pain if there weren't something potentially dangerous going on in my body | 1 | 2 | 3 | 4 |
| 12. Although my condition is painful, I would be better off if I were physically active | 1 | 2 | 3 | 4 |
| 13. Pain lets me know when to stop exercising so that I don't injure myself | 1 | 2 | 3 | 4 |
| 14. It's really not safe for a person with a condition like mine to be physically active | 1 | 2 | 3 | 4 |
| 15. I can't do all the things normal people do because it's too easy for me to get injured | 1 | 2 | 3 | 4 |
| 16. Even though something is causing me a lot of pain, I don't think it's actually dangerous | 1 | 2 | 3 | 4 |
| 17. No one should have to exercise when he/she is in pain | 1 | 2 | 3 | 4 |

Scoring Information Tampa Scale for Kinesiophobia (Miller et al., 1991)

A total score is calculated after inversion of the individual scores of items 4, 8, 12 and 16.


### 2000 IKDC SUBJECTIVE KNEE EVALUATION FORM

| Nar | ne: | | | | | Date | e: | | | | Physician: |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Dat | e of Inj | ury: | | | | | | | | | |
| SYI | MPTON | MS*: | | | | | | | | | |
| fur | rade synction wities a | ithout s | ignifica | _ | • | | | • | • | could<br>rforming | |
| 1. V | Vhat is t | he high | est leve | l of acti | vity tha | t you ca | n perfo | rm with | nout sig | nificant kı | nee pain? |
| S<br>M<br>I | Very street<br>Strenuou<br>Moderate<br>Light act<br>Jnable to | s activi<br>e activit | ties like<br>ties like<br>like wal | heavy<br>modera | physica<br>nte phys | l work, ical wo | skiing o | or tenni | s<br>ogging | | |
| 2. D | ouring th | ne <u>past</u> 4 | 4 weeks | , or sinc | e your | injury, l | now ofte | en have | you ha | d pain? | |
| 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | |
| Nev | er | | | | | | | | | Constar | nt |
| 3. If | f you ha | ve pain, | , how se | evere is | it? | | | | | | |
| 0 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | |
| No | pain | | | | | | | | Worse | pain imag | ginable |
| 4. D | ouring th | ne past 4 | 4 weeks | , or sinc | e your i | injury, 1 | now stif | f or sw | ollen w | as your kn | iee |


| Mildly |
|---|
| Moderately |
| Very |
| Extremely |
| 5. What is the highest level of activity you can perform without significant swelling in your |
| knee? |
| Very strenuous activities like jumping or pivoting as in basketball or soccer |
| Strenuous activities like heavy physical work, skiing or tennis |
| Moderate activities like moderate physical work, running or jogging |
| Light activities like walking, housework, or yard work |
| Unable to perform any of the above activities due to giving way of the knee |
| 6. During the past 4 weeks, or since your injury, did your knee lock or catch? |
| Yes No |
| 7. What is the highest level of activity you can perform without significant giving way in your |
| knee? |
| Very strenuous activities like jumping or pivoting as in basketball or soccer |
| Strenuous activities like heavy physical work, skiing or tennis |
| Moderate activities like moderate physical work, running or jogging |
| Light activities like walking, housework, or yard work |
| Unable to perform any of the above activities due to giving way of the knee |
| SPORTS ACTIVITIES: |
| 8. What is the highest level of activity you can participate in on a regular basis? |

Not at all

Version: 1.0 Version Date: 10NOV2021

Very strenuous activities like jumping or pivoting as in basketball or soccer

Strenuous activities like heavy physical work, skiing or tennis

Moderate activities like moderate physical work, running or jogging

Light activities like walking, housework, or yard work

Unable to perform any of the above activities due to giving way of the knee

9. How does your knee affect your ability to:

| | | Not<br>difficult<br>at all | Minimall<br>y<br>difficult | Moderate<br>ly<br>Difficult | Extremel<br>y<br>difficult | Unable<br>to do |
|---|---|---|---|---|---|---|
| A. | Go up stairs | 0 | 0 | 0 | 0 | 0 |
| B. | Go down stairs | 0 | 0 | 0 | 0 | 0 |
| C. | Kneel on the front of your knee | 0 | О | 0 | 0 | 0 |
| D. | Squat | 0 | 0 | 0 | 0 | 0 |
| E. | Sit with your knee bent | 0 | 0 | 0 | 0 | 0 |
| F. | Rise from a chair | 0 | 0 | 0 | 0 | 0 |
| G. | Run straight ahead | 0 | 0 | 0 | 0 | 0 |


| Н. | | and la | and on y | rour | 0 | 0 | | 0 | , | 0 | 0 |
|---|---|---|---|---|---|---|---|---|---|---|---|
| I. | Stop | and sta | art quicl | dy | 0 | 0 | | 0 | | 0 | 0 |
| FUN | CTION: | | | | | | | | | | |
| norm | ities whi | llent fu<br>ich ma | unction a<br>y includ<br>OR TO Y | and 0 b<br>le sport<br>YOUR | eing the in | ability<br>JURY: | | | | ) with 10 bei<br>our usual dai | ily |
| Could | n't perform ( | daily | | | | | | | | No limitation | s in daily activities |
| CUR | RENT I | FUNC | ΓΙΟΝ Ο | F YOU | JR KNEE: | | | | | | |
| 0 | | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 |
| Canno<br>activit | ot perform da | aily | | | | | | | | No limitatio | n in daily activities |

Version: 1.0 Version Date: 10NOV2021

## Single Leg Squat Scoring

| Grade | Hip and Knee Criteria |
|---|---|
| Excellent | Hip flexion greater than 65°, hip abduction / adduction less than 10°, knee valgus / varus less than 10° |
| Good | Any of the above 2 criteria are met |
| Fair | Any 1 of the above criteria are met |
| Poor | None of the criteria are met or the athlete losses balance or falls |

Figure 1. Single leg squat - Scoring Criteria for movements of closed chain limb

| Single Leg Squat Assessment | | Left | Right |
|---|---|---|---|
| Foot | Foot Flattens | yes/no | yes/no |
| Knee | Positioning/Valgus | Moves Inward Moves Outward | Moves Inward Moves Outward |
| Pelvic Plane | Excessive Tilt (Ant/Post) | yes/no | yes/no |
| Stance/Stability | Stability: Noticeable instability | yes/no | yes/no |
| Pain | Verbal report of pain | yes/no | yes/no |

Table 1. Single leg squat assessment
